CLINICAL TRIAL: NCT01044498
Title: An Open-label, Multi-center, One Sequence Cross-over Drug Interaction Study to Investigate the Effect of Tocilizumab (TCZ, RO4877533) on the Pharmacokinetics and Pharmacodynamics of an Oral Contraceptive (OC) in Female Patients With Active Rheumatoid Arthritis (RA)
Brief Title: A Study of Tocilizumab in Combination With an Oral Contraceptive in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP22775
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (2):
- Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) (Experimental): Patients with rheumatoid arthritis received Ortho-Novum® 1/35 daily on Days 1-21 of 3 consecutive 28-day cycles. On the first day of Cycle 2, patients received tocilizumab 8 mg/kg administered intravenously.
  Interventions: Drug: Tocilizumab; Drug: Ortho-Novum® 1/35
- Ortho-Novum® 1/35 (Group 2) (Other): Healthy volunteers received Ortho-Novum® 1/35 tablets daily on Days 1-21 of one 28-day cycle.
  Interventions: Drug: Ortho-Novum® 1/35

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 8 mg/kg was administered in a single 1-hour infusion on Day 1 of Cycle 2.
  Other Names: RoActemra; Actemra
  Arms: Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1)
Drug: Ortho-Novum® 1/35 — Each Ortho-Novum® 1/35 tablet contained 1 mg of norethindrone and 0.035 mg of ethinyl estradiol.

SUMMARY:
This open-label, randomized, cross-over study evaluated the effect of tocilizumab (TCZ) on the pharmacokinetics and pharmacodynamics of a common oral contraceptive (OC) in female patients with active rheumatoid arthritis (RA) and in healthy female volunteers of child bearing age. The RA patients received OC in combination with TCZ, whereas the healthy volunteers received OC only. The RA patients received OC in 3 cycles of 21 days each; TCZ 8 mg/kg was administered once as an intravenous infusion on the first day of Cycle 2. The healthy volunteers received OC for only one 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with child bearing potential, 18-44 years of age.
* Rheumatoid arthritis (RA) for over 6 months duration.
* On oral contraceptive without interruption for at least 3 months with normal cycle control.
* Treatment with disease-modifying anth-rheumatic drugs (DMARD) for at least 12 weeks prior to study start.
* Body weight < 150 kg.

Exclusion Criteria:

* Functional class IV rheumatoid arthritis (American College of Rheumatology [ACR] classification).
* History of amenorrhea (unrelated to pregnancy).
* History or current inflammatory joint disease other than RA.
* Rheumatic autoimmune disease other than RA.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (6):
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Ormond Beach, Florida
  - Port Orange, Florida
  - Duncansville, Pennsylvania
  - San Antonio, Texas

REFERENCES:
- [Derived] Zhang X, Rowell L, Fettner S, Lau C, Teuber D. Assessment of disease-drug-drug interaction between single-dose tocilizumab and oral contraceptives in women with active rheumatoid arthritis. Int J Clin Pharmacol Ther. 2014 Jan;52(1):27-38. doi: 10.5414/CP201951. PMID 24161161

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) | Ortho-Novum® 1/35 (Group 2)
Started | 23 | 23
Completed | 20 | 21
Not Completed | 3 | 2
Not completed — Withdrew consent | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) | Ortho-Novum® 1/35 (Group 2) | Total
Number analyzed (Participants) | 23 | 23 | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 35.8 (7.66) | 25.7 (5.04) | 30.7 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Serum Progesterone Level
Description: Blood samples were collected prior to the administration of Ortho-Novum® 1/35 on Day 21 of each cycle. Serum levels of progesterone were quantitatively determined using the ADVIA Centaur and ADVIA Centaur XP systems (Siemens Healthcare Diagnostics Inc., Tarrytown, NY, USA). The assay was a competitive immunoassay using direct chemiluminescent technology.
Time Frame: Day 21 of Cycles 1-3 for Group 1 and Day 21 of Cycle 1 for Group 2
Population: Pharmacokinetic (PK) and pharmacodynamic (PD) population: All patients enrolled in the study who had at least 1 evaluable PK or PD sample reading. Blood samples were not available for all patients at all time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) | Ortho-Novum® 1/35 (Group 2)
Number analyzed (Participants) | 22 | 16
ng/mL
  Cycle 1 (n=22, 16) | 0.21 (0.07) | 0.57 (0.39)
  Cycle 2 (n=19, NA) | 0.22 (0.10) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3 (n=18, NA) | 0.19 (0.00) | NA (NA) — There was only 1 cycle for Group 2.

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ethinyl Estradiol and Norethindrone
Description: Blood samples were collected prior to and at 0.5, 1, 1.5, 2, 3, 5, 8, 12 and 24 hours after administration of Ortho-Novum® 1/35 on Day 7 of each cycle. The concentrations of ethinyl estradiol and norethindrone were determined in human heparinized plasma according to a validated gas chromatography coupled to mass spectrometry (GC-MS) method. The maximum observed plasma concentration (Cmax) was derived from the plasma concentrations using a non-compartmental method with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: Day 7 of Cycles 1-3 for Group 1 and Day 7 of Cycle 1 for Group 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) | Ortho-Novum® 1/35 (Group 2)
Number analyzed (Participants) | 22 | 21
pg/mL
  Cycle 1, ethinyl estradiol, N=22,21 | 183 (86.2) | 157 (53.3)
  Cycle 2, ethinyl estradiol, N=18,NA | 163 (71.4) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, ethinyl estradiol, N=18,NA | 177 (104.2) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 1, norethindrone, N=22,21 | 13396 (4687.9) | 18943 (5570.6)
  Cycle 2, norethindrone, N=18,NA | 14747 (4215.8) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, norethindrone, N=18,NA | 15772 (4863.4) | NA (NA) — There was only 1 cycle for Group 2.

3. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Ethinyl Estradiol and Norethindrone
Description: Blood samples were collected prior to and at 0.5, 1, 1.5, 2, 3, 5, 8, 12 and 24 hours after administration of Ortho-Novum® 1/35 on Day 7 of each cycle. The concentrations of ethinyl estradiol and norethindrone were determined in human heparinized plasma according to a validated gas chromatography coupled to mass spectrometry (GC-MS) method. The time to reach the maximum plasma concentration (Tmax) was derived from the plasma concentrations using a non-compartmental method with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: Day 7 of Cycles 1-3 for Group 1 and Day 7 of Cycle 1 for Group 2
Population: Pharmacokinetic (PK) and pharmacodynamic (PD) population: All patients enrolled in the study who had at least 1 evaluable PK or PD sample reading.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) | Ortho-Novum® 1/35 (Group 2)
Number analyzed (Participants) | 22 | 21
hr
  Cycle 1, ethinyl estradiol | 1.42 (0.68) | 1.28 (0.54)
  Cycle 2, ethinyl estradiol | 1.90 (2.69) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, ethinyl estradiol | 1.58 (0.73) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 1, norethindrone | 1.33 (0.73) | 1.02 (0.47)
  Cycle 2, norethindrone | 1.82 (1.59) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, norethindrone | 1.30 (0.46) | NA (NA) — There was only 1 cycle for Group 2.

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC0-24) of Ethinyl Estradiol and Norethindrone
Description: Blood samples were collected prior to and at 0.5, 1, 1.5, 2, 3, 5, 8, 12 and 24 hours after administration of Ortho-Novum® 1/35 on Day 7 of each cycle. The concentrations of ethinyl estradiol and norethindrone were determined in human heparinized plasma according to a validated gas chromatography coupled to mass spectrometry (GC-MS) method. The area under the plasma concentration-time curve from 0 to 24 hours (AUC0-24) was derived from the plasma concentrations using a non-compartmental method and computed using the linear trapezoidal rule with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: Day 7 of Cycles 1-3 for Group 1 and Day 7 of Cycle 1 for Group 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg•hr/mL
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) | Ortho-Novum® 1/35 (Group 2)
Number analyzed (Participants) | 22 | 21
pg•hr/mL
  Cycle 1, ethinyl estradiol | 1387 (453) | 1389 (502)
  Cycle 2, ethinyl estradiol | 1409 (552) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, ethinyl estradiol | 1455 (487) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 1, norethindrone | 108513 (39795) | 128975 (53276)
  Cycle 2, norethindrone | 120505 (43285) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, norethindrone | 121667 (47828) | NA (NA) — There was only 1 cycle for Group 2.

5. Secondary Outcome: Terminal Half-life (t½) of Ethinyl Estradiol and Norethindrone
Description: Blood samples were collected prior to and at 0.5, 1, 1.5, 2, 3, 5, 8, 12 and 24 hours after administration of Ortho-Novum® 1/35 on Day 7 of each cycle. The concentrations of ethinyl estradiol and norethindrone were determined in human heparinized plasma according to a validated gas chromatography coupled to mass spectrometry (GC-MS) method. The terminal half-life (t½) was derived from the plasma concentrations using a non-compartmental method with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: Day 7 of Cycles 1-3 for Group 1 and Day 7 of Cycle 1 for Group 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) | Ortho-Novum® 1/35 (Group 2)
Number analyzed (Participants) | 22 | 21
hr
  Cycle 1, ethinyl estradiol | 14.71 (9.10) | 17.05 (9.71)
  Cycle 2, ethinyl estradiol | 14.70 (7.47) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, ethinyl estradiol | 15.24 (6.78) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 1, norethindrone | 12.18 (4.49) | 11.54 (4.20)
  Cycle 2, norethindrone | 13.48 (3.69) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, norethindrone | 16.14 (10.97) | NA (NA) — There was only 1 cycle for Group 2.

6. Secondary Outcome: Apparent Oral Clearance (CL/F) of Ethinyl Estradiol and Norethindrone
Description: Blood samples were collected prior to and at 0.5, 1, 1.5, 2, 3, 5, 8, 12 and 24 hours after administration of Ortho-Novum® 1/35 on Day 7 of each cycle. The concentrations of ethinyl estradiol and norethindrone were determined in human heparinized plasma according to a validated gas chromatography coupled to mass spectrometry (GC-MS) method. The apparent oral clearance (CL/F) was derived from the plasma concentrations using a non-compartmental method and computed as dose/AUC0-24 with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: Day 7 of Cycles 1-3 for Group 1 and Day 7 of Cycle 1 for Group 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) | Ortho-Novum® 1/35 (Group 2)
Number analyzed (Participants) | 22 | 21
mL/hr
  Cycle 1, ethinyl estradiol | 28.49 (11.40) | 28.64 (11.06)
  Cycle 2, ethinyl estradiol | 29.23 (12.88) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, ethinyl estradiol | 26.86 (9.38) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 1, norethindrone | 10.40 (3.59) | 9.05 (3.71)
  Cycle 2, norethindrone | 9.45 (3.59) | NA (NA) — There was only 1 cycle for Group 2.
  Cycle 3, norethindrone | 9.53 (3.72) | NA (NA) — There was only 1 cycle for Group 2.

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Tocilizumab
Description: Blood samples were collected pre-dose and at the end of infusion of tocilizumab on Day 1 of Cycle 2. Additional blood samples were collected on Days 2, 3, 5, 7, 12, 14, 21 of Cycle 2, and Days 1, 7, and 21 of Cycle 3. The concentration of tocilizumab was determined in serum samples using a validated enzyme-linked immunosorbent assay (ELISA). The maximum observed plasma concentration (Cmax) was derived from the serum concentrations using a non-compartmental method with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: From Day 1 of Cycle 2 to Day 21 of Cycle 3 for Group 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1)
Number analyzed (Participants) | 20
µg/mL | 204 (63.4)

8. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of Tocilizumab
Description: Blood samples were collected pre-dose and at the end of infusion of tocilizumab on Day 1 of Cycle 2. Additional blood samples were collected on Days 2, 3, 5, 7, 12, 14, 21 of Cycle 2, and Days 1, 7, and 21 of Cycle 3. The concentration of tocilizumab was determined in serum samples using a validated ELISA. The time to reach maximum serum concentration was derived from the serum concentrations using a non-compartmental method with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: From Day 1 of Cycle 2 to Day 21 of Cycle 3 for Group 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1)
Number analyzed (Participants) | 20
hr | 4.41 (8.39)

9. Secondary Outcome: Area Under the Serum Concentration-time Curve From 0 to Infinity (AUCinf) of Tocilizumab
Description: Blood samples were collected pre-dose and at the end of infusion of tocilizumab on Day 1 of Cycle 2. Additional blood samples were collected on Days 2, 3, 5, 7, 12, 14, 21 of Cycle 2, and Days 1, 7, and 21 of Cycle 3. The concentration of tocilizumab was determined in serum samples using a validated ELISA. The area under the serum concentration-time curve from 0 to infinity (AUCinf) was derived from the serum concentrations using a non-compartmental method with the software WinNonlin Enterprise version 5.2 (or above). AUCinf was computed using the linear trapezoidal rule to tlast plus Clast/Kel, where tlast is the time of the last measurable concentration, Clast is the last measurable concentration, and Kel is the apparent elimination rate, computed as the magnitude of the slope from the log-linear regression of the apparent terminal elimination phase of the serum concentration-versus-time curve.
Time Frame: From Day 1 of Cycle 2 to Day 21 of Cycle 3 for Group 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg•hr/mL
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1)
Number analyzed (Participants) | 20
µg•hr/mL | 35038 (8324)

10. Secondary Outcome: Terminal Half-life (t½) of Tocilizumab
Description: Blood samples were collected pre-dose and at the end of infusion of tocilizumab on Day 1 of Cycle 2. Additional blood samples were collected on Days 2, 3, 5, 7, 12, 14, 21 of Cycle 2, and Days 1, 7, and 21 of Cycle 3. The concentration of tocilizumab was determined in serum samples using a validated ELISA. The terminal half-life (t½) was derived from the serum concentrations using a non-compartmental method with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: From Day 1 of Cycle 2 to Day 21 of Cycle 3 for Group 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1)
Number analyzed (Participants) | 20
hr | 145.92 (57.69)

11. Secondary Outcome: Clearance (CL) of Tocilizumab
Description: Blood samples were collected pre-dose and at the end of infusion of tocilizumab on Day 1 of Cycle 2. Additional blood samples were collected on Days 2, 3, 5, 7, 12, 14, 21 of Cycle 2, and Days 1, 7, and 21 of Cycle 3. The concentration of tocilizumab was determined in serum samples using a validated ELISA. Clearance (CL), computed as dose/AUCinf, was derived from the serum concentrations using a non-compartmental method with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: From Day 1 of Cycle 2 to Day 21 of Cycle 3 for Group 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1)
Number analyzed (Participants) | 20
mL/hr | 17.51 (4.59)

12. Secondary Outcome: Apparent Volume of Distribution (Vz) of Tocilizumab
Description: Blood samples were collected pre-dose and at the end of infusion of tocilizumab on Day 1 of Cycle 2. Additional blood samples were collected on Days 2, 3, 5, 7, 12, 14, 21 of Cycle 2, and Days 1, 7, and 21 of Cycle 3. The concentration of tocilizumab was determined in serum samples using a validated ELISA. The apparent volume of distribution (Vz), computed as CL/Kel where CL is clearance and Kel is the apparent elimination rate, was derived from the serum concentrations using a non-compartmental method with the software WinNonlin Enterprise version 5.2 (or above).
Time Frame: From Day 1 of Cycle 2 to Day 21 of Cycle 3 for Group 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1)
Number analyzed (Participants) | 20
L | 3.60 (1.37)

13. Secondary Outcome: Serum Soluble Interleukin-6 Receptor (sIL-6R) Level
Description: Blood samples were collected pre-dose and at the end of infusion of tocilizumab on Day 1 of Cycle 2. Additional blood samples were collected on Days 2, 3, 5, 7, 12, 14, and 21 of Cycle 2, and Days 1, 7, and 21 of Cycle 3. Serum levels of soluble interleukin-6 receptor were analyzed using a validated ELISA.
Time Frame: From Day 1 of Cycle 2 to Day 21 of Cycle 3 for Group 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1)
Number analyzed (Participants) | 21
ng/mL
  Cycle 2, Day 1 | 38.5 (10.3)
  Cycle 2, Day 2 | 100.6 (23.7)
  Cycle 2, Day 3 | 162.5 (52.8)
  Cycle 2, Day 5 | 249.1 (68.2)
  Cycle 2, Day 7 | 312.9 (63.6)
  Cycle 2, Day 12 | 425.1 (78.0)
  Cycle 2, Day 14 | 476.2 (89.1)
  Cycle 2, Day 21 | 503.2 (131.8)
  Cycle 3, Day 1 | 534.9 (169.4)
  Cycle 3, Day 7 | 387.3 (188.0)
  Cycle 3, Day 21 | 45.7 (12.4)

14. Secondary Outcome: Serum C-reactive Protein (CRP) Level
Description: Blood samples were collected pre-dose of tocilizumab infusion on Day 1 of Cycle 2 and on Days 2, 3, 5, 7, 12, 14, and 21 of Cycle 2, and on Days 1, 7, and 21 of Cycle 3. Serum levels of C-reactive protein were measured by the Tina-quant CRP (latex) high-sensitivity Roche Immunoturbidimetric method.
Time Frame: From Day 1 of Cycle 2 to Day 21 of Cycle 3 for Group 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1)
Number analyzed (Participants) | 21
mg/L
  Cycle 2, Day 1 | 16.86 (21.55)
  Cycle 2, Day 2 | 12.76 (16.07)
  Cycle 2, Day 3 | 7.53 (12.61)
  Cycle 2, Day 5 | 4.62 (12.47)
  Cycle 2, Day 7 | 3.90 (12.42)
  Cycle 2, Day 12 | 3.95 (13.22)
  Cycle 2, Day 14 | 3.92 (13.03)
  Cycle 2, Day 21 | 3.97 (12.95)
  Cycle 3, Day 1 | 3.74 (11.96)
  Cycle 3, Day 7 | 8.11 (13.62)
  Cycle 3, Day 21 | 12.37 (9.42)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of signing informed consent through the follow-up visit.
Description: The safety analysis population included all subjects who received at least 1 study dose and had at least 1 post-dose safety assessment.
Arm/Group | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) | Ortho-Novum® 1/35 (Group 2)
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/23
Other Adverse Events (participants affected / at risk) | 12/23 | 4/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) (N=23) | Ortho-Novum® 1/35 (Group 2) (N=23)
Hypersensitivity (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg + Ortho-Novum® 1/35 (Group 1) (N=23) | Ortho-Novum® 1/35 (Group 2) (N=23)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Headache (Nervous system disorders) | 3 | 0
LFT abnormal (Investigations) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Systolic hypertension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.